CLINICAL TRIAL: NCT01416779
Title: Finding Balance: The Experience of Hope for Bereaved Caregivers of Palliative Cancer Patients
Brief Title: A Finding Balance Writing Intervention for Older Bereaved Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Principal Investigator, Lorraine Holtslander, Associate Professor, University of Saskatchewan
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 08-154
Record Dates: First submitted 2011-02-07; First posted 2011-08-15 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Grief
Keywords: Writing Intervention; Bereaved Caregivers; Older Adults; hope; inventory of daily widowed life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Writing Group (Experimental): This group will receive the writing intervention.
  Interventions: Behavioral: Writing Intervention
- No Intervention (No Intervention): Non Writing Group

INTERVENTIONS:
Behavioral: Writing Intervention — Finding Balance Writing Intervention
  Arms: Writing Group

SUMMARY:
The overall purpose of this study is to develop and pilot-test a theory-based psychosocial supportive "finding balance" intervention for older, bereaved spousal caregivers of a palliative cancer patient.

DETAILED DESCRIPTION:
Research devoted to determining the efficacy of bereavement interventions remains a top priority. The development of theory-based, acceptable and feasible psychosocial interventions would begin to address the needs of family caregivers. A prominent theory of coping with bereavement, Stroebe and Schut's Dual Process Model, describes oscillation between loss-oriented and restoration-oriented coping; having a balance between these processes predicted more positive outcomes for older bereaved spouses. Similarly, the process of "finding balance" emerged as a first step in the search for new hope in the PI's grounded theory research with older bereaved family caregivers. They described the importance and difficulty of "finding balance" as they recovered from caregiving and struggled to find a new meaning and purpose for their lives after the loss of a spouse to cancer. An intervention focused on "finding balance" provides an innovative and promising approach to guiding the development of a theory-based psychosocial intervention for family caregivers who become bereaved. In clinical work a highly focused writing intervention has shown important benefits (personal communication, Dr. Robert Neimeyer, March 4, 2009). A validated tool to measure the effectiveness of an intervention to find balance does not exist, however valid existing measures of hope, grief, and an inventory of balance based on the Dual Process Model will be used as proxies. Therefore, the overall purpose of this study is to develop and pilot-test a theory-based psychosocial supportive "finding balance" intervention for older, bereaved spousal caregivers of a palliative cancer patient.

ELIGIBILITY:
Inclusion Criteria:

* women and men, ages 60 and over, who previously resided with and provided care for a spouse with terminal cancer who died within the last year, English speaking, and freely consenting to be involved in the study.

Exclusion Criteria:

* will be those cognitively impaired, non-autonomous, or not able to give a free and informed consent, as determined by the registered nurse research assistant on initial contact.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Grief | 2 weeks
  Herth Hope Index, Hogan Grief Scale, Inventory of Daily Widowed Life, Finding Balance Scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Holtslander LF, Bally JM, Steeves ML. Walking a fine line: an exploration of the experience of finding balance for older persons bereaved after caregiving for a spouse with advanced cancer. Eur J Oncol Nurs. 2011 Jul;15(3):254-9. doi: 10.1016/j.ejon.2010.12.004. Epub 2011 Jan 17. PMID 21247803